CLINICAL TRIAL: NCT01963416
Title: A Randomized Controlled, Crossover in Design, Double Blind Clinical Trial Investigating the Effects of Whole Versus Processed Fruit Consumption on Risk Factors for Chronic Disease and Performance Indicators.
Brief Title: Effects of Fruit Consumption on Risk Factors of Chronic Disease
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Reading (Other)
Collaborators: PepsiCo Global R&D (Industry)
Responsible Party: Principal Investigator, Jeremy Paul Edward Spencer, Professor of Nutritional Medicine, University of Reading
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: UOR-0001
Record Dates: First submitted 2013-10-10; First posted 2013-10-16 (Estimated); Last update posted 2013-10-16 (Estimated); Status verified 2013-10

CONDITIONS: Vascular Stiffness

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Control (Placebo Comparator): macro- and micro-nutrient matched control (240 ml)
  Interventions: Dietary Supplement: macro- and micro-nutrient matched control (240 ml)
- Orange juice (Experimental): commercial orange juice (240 ml)
  Interventions: Dietary Supplement: Orange juice
- whole orange (Experimental): whole orange fruit (240 ml)
  Interventions: Dietary Supplement: whole orange fruit
- processed whole orange (Experimental): processed whole orange (240 ml)
  Interventions: Dietary Supplement: Processed whole orange

INTERVENTIONS:
Dietary Supplement: macro- and micro-nutrient matched control (240 ml)
  Arms: Control
Dietary Supplement: Orange juice
  Arms: Orange juice
Dietary Supplement: whole orange fruit
  Arms: whole orange
Dietary Supplement: Processed whole orange
  Arms: processed whole orange

SUMMARY:
Acute, randomized, placebo controlled, double blind, postprandial crossover study in male subjects. 4 intervention arms consisting of control, orange juice, whole orange, and processed whole orange to determine the effect of the interventions on the primary measure of flow mediated dilatation (FMD) and additional biomarkers of health. The study will also identify and quantify the main micronutrients and phytochemicals in each of the products and will identify and quantify the main micronutrients and phytochemicals and their metabolites in the subjects' plasma and/or urine. A subset of the study population (n=24) will be invited to participate in an additional arm of the main study which is summarised below.

ELIGIBILITY:
Inclusion Criteria:

* Males due to potential hormonal fluctuations in female subjects
* Aged 30-65years
* Fasting total cholesterol in the upper half of the normal range (6.0-8.0 mmol/l) or triacylglycerol >0.8 mmol/l or a BMI 25-32 kg/m2.
* Not having suffered a myocardial infarction/stroke in the past 12 months
* Not diabetic (diagnosed or fasting glucose > 7 mmol/l) or suffer from other endocrine disorders
* Not suffering from renal or bowel disease or have a history of choleostatic liver or pancreatitis
* Not on drug treatment for hyperlipidaemia, hypertension, inflammation or hypercoagulation
* No history of alcohol misuse
* Not planning or on a weight reducing regime
* Not taking any fish oil, fatty acid or vitamin and mineral supplements
* Non smokers
* Not suffering from depression as indicated by the Brief Symptom Inventory (Appendix 11).
* Not suffering from mild cognitive impairment or dementia according to the MMSE (score ≥ 25).

Exclusion Criteria:

* Females
* Medication for hypertension, hyperlipidaemia, inflammation or hypercoagulation

  * Hypertension - ACE Inhibitors (e.g. Captopril, Cilazapril), Angiotensin Receptor Blockers (Valsartan), Calcium Channel Blockers (Amlodipine, Nicardipine), Diuretics (Chlortalidone) or Beta blockers (Sotalol, Bisoprolol).
  * Cholesterol lowering (Pravastatin, Simuvustatin)
  * Anticoagulants (Warfarin)
  * Inflammation - NSAID's (Tiaprofenic acid, Sulindac, Ibuprofen), Corticosteroids(Betamethasone)
* Strict vegetarians
* Smokers
* Those on or planning a weight reducing regime
* Blood glucose, haemaglobin or liver enzymes outside of the normal range
* Unable to consume study meals
* Those suffering from depression as indicated by the Brief Symptom Inventory (Appendix 11).
* Those suffering from mild cognitive impairment or dementia as indicated by the MMSE (score < 25).

Ages: 30 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2012-06; Primary Completion 2012-12 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Flow mediated dilation | change in Flow Mediated Dilation response between baseline and 6 hours

SECONDARY OUTCOMES:
Postprandial plasma glucose | change in glucose from baseline to 2 hours
Postprandial insulin | change from baseline to 2 hours
global cognitive function | change from baseline to 6 hours
Blood pressure | change from baseline to 6 hours
postprandial non-esterified fatty acids | change from baseline to 6 hours
Postprandial triacylglycerol | change from baseline to 6 hours
total HDL/LDL | change from baseline to 6 hours
Inflammatory status (IL1-beta; IL2; IL6; IL10; IFN-gamma; TNF-alpha; CRP) | change from baseline to 6 hours
LDL oxidation | change from baseline to 6h

OTHER OUTCOMES:
Plasma flavanone metabolites | change from baseline to 6 hours

CONTACTS AND LOCATIONS:
Locations (1):
- University of Reading, Reading, Berkshire, United Kingdom

REFERENCES:
- [Derived] Dong H, Rendeiro C, Kristek A, Sargent LJ, Saunders C, Harkness L, Rowland I, Jackson KG, Spencer JP, Lovegrove JA. Addition of Orange Pomace to Orange Juice Attenuates the Increases in Peak Glucose and Insulin Concentrations after Sequential Meal Ingestion in Men with Elevated Cardiometabolic Risk. J Nutr. 2016 Jun;146(6):1197-203. doi: 10.3945/jn.115.226001. Epub 2016 May 11. PMID 27170728